CLINICAL TRIAL: NCT03373422
Title: A Randomized, Placebo-controlled, Double-blind, Parallel-group, Multi-center, Exploratory Dose-response Study to Assess the Efficacy and Safety of Different Oral Doses of BAY1128688 in Women With Symptomatic Endometriosis Over a 12-week Treatment Period
Brief Title: A Study to Test Whether Study Drug BAY1128688 Brings Pain Relief to Women With Endometriosis and if so to Get a First Idea Which Dose(s) Work Best
Acronym: AKRENDO1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study BAY1128688/17472 (AKRENDO 1) was terminated early on 20 July 2018 due to hepatotoxicity
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17472; 2017-000244-18 (EudraCT Number)
Record Dates: First submitted 2017-11-23; First posted 2017-12-14 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — BAY1128688

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- BAY1128688 (dose 1) (Experimental): One BAY1128688 tablet (lowest dose) in the morning, one placebo tablet in the evening
  Interventions: Drug: BAY1128688; Drug: Placebo
- BAY1128688 (dose 2) (Experimental): One BAY1128688 tablet (first intermediate dose) in the morning, one placebo tablet in the evening
  Interventions: Drug: BAY1128688; Drug: Placebo
- BAY1128688 (dose 3) (Experimental): One BAY1128688 tablet (second intermediate dose) in the morning, one placebo tablet in the evening
  Interventions: Drug: BAY1128688; Drug: Placebo
- BAY1128688 (dose 4) (Experimental): One BAY1128688 tablet (second intermediate dose) in the morning and one in the evening
  Interventions: Drug: BAY1128688
- BAY1128688 (dose 5) (Experimental): One BAY1128688 tablet (highest dose) in the morning and one in the evening
  Interventions: Drug: BAY1128688
- Placebo (Placebo Comparator): One placebo tablet in the morning and one in the evening
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY1128688 — Various dosing OD (once daily) and BID (twice daily)
  Arms: BAY1128688 (dose 1); BAY1128688 (dose 2); BAY1128688 (dose 3); BAY1128688 (dose 4); BAY1128688 (dose 5)
Drug: Placebo — Matching placebo tablets
  Arms: BAY1128688 (dose 1); BAY1128688 (dose 2); BAY1128688 (dose 3); Placebo

SUMMARY:
Purpose of the study is to test whether study drug BAY1128688 brings relief for pain to women with endometriosis and if so to get a first impression which dose(s) work best.

ELIGIBILITY:
Inclusion Criteria:

* Women of at least 18 years of age at the time of signing of informed consent
* Women with endometriosis confirmed by at least one of the two criteria:

  * surgery within the last 10 years
  * imaging within the last 12 months
* moderate to severe pelvic pain which will be assessed over a period of 28 days
* Willingness to use only ibuprofen as rescue pain medication for endometriosis-associated pelvic pain
* Willingness to use non-hormonal barrier method for contraception (here spermicide-coated condoms) from screening visit until the end of the study (unless adequate contraception is achieved by vasectomy of the partner or use of copper intrauterine device [IUD] or commitment to abstinence) and refrain from using hormonal contraception

Exclusion Criteria:

* Pregnancy or lactation (more than three months since delivery, abortion, or lactation before start of treatment) AND no wish for pregnancy during the study
* Altered bilirubin metabolism and liver function at Visit 1
* Requirement to use pain medications for reasons other than endometriosis
* Contraindications to using ibuprofen
* Signs of hyperandrogenism
* Absence of menstrual cycles and/or abnormal vaginal/genital bleeding
* History of hysterectomy, tubal-ligation or bilateral ovariectomy
* Uncontrolled thyroid disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Absolute change in mean pain of the 7 days with worst EAPP comparing the 28-day baseline cycle (baseline period of daily pain recordings) to the 28-day end of treatment cycle (daily pain recordings during the last 28 days of the treatment period) | 12 weeks
  EAPP: endometriosis-associated pelvic pain, measured on the NRS (Numerical Rating Scale) by item 1 of the ESD (Endometriosis Symptom Diary)

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (67):
- Austria (4):
  - Medizinische Universität Graz, Graz, Styria
  - Kepler Universitätsklinikum, Linz, Upper Austria
  - Landeskrankenhaus - Universitätskliniken Innsbruck, Innsbruck
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
- Belgium (4):
  - AZ Jan Palfijn Gent, Ghent, Oost-Vlaanderen
  - CU Saint-Luc/UZ St-Luc, Bruxelles - Brussel
  - Ziekenhuis Oost-Limburg, Genk
  - CHU de Tivoli, La Louvière
- Czechia (6):
  - Gynekologie MEDA s.r.o., Brno
  - GYN-F s.r.o., Hradec Králové
  - G-Centrum Olomouc s.r.o. Dr. Skrivanek, Olomouc
  - GynCare MUDr. Michael Svec s.r.o., Pilsen
  - Centrum gynekologicke rehabilitace, Písek
  - Dr. Smrhova-Kovacs, Tábor
- Denmark (2):
  - Aarhus Universitetshospital, Skejby, Aarhus N
  - H:S Rigshospitalet, København Ø
- Finland (4):
  - HUS / Naistenklinikka, Helsinki
  - Keski-Suomen keskussairaala, Jyväskylä
  - Lääkäriasema Cantti Oy, Kuopio
  - Lääkärikeskus Gyneko, Oulu
- France (2):
  - Centre Hospitalier Universitaire - Angers, Angers
  - Cochin - Paris, Paris
- Germany (10):
  - Vincentius-Diakonissen-Kliniken gAG, Karlsruhe, Baden-Wurttemberg
  - Praxisklinik am Rosengarten, Mannheim, Baden-Wurttemberg
  - Klinikum rechts der Isar, München, Bavaria
  - Praxis Hr. Dr. A. Gerick, Aachen, North Rhine-Westphalia
  - Praxis Hr. Dr. S. Fiedler, Aachen, North Rhine-Westphalia
  - Frauenarztpraxis Dr. Wolfgang Clemens, Stolberg, North Rhine-Westphalia
  - Praxis f. Gynäkologie und Geburtshilfe, Bernburg, Saxony-Anhalt
  - Frauenarztpraxis Dr. Wetzel, Blankenburg, Saxony-Anhalt
  - Praxis Hr. Prof. Dr. A. Ebert, Berlin
  - Charité Campus Benjamin Franklin (CBF), Berlin
- Hungary (7):
  - Semmelweis University, Budapest
  - Bajcsy Zsilinszky Korhaz-Rendelointezet, Budapest
  - Robert Karoly Magankorhaz, Budapest
  - NAP - Rendelo, Private Clinic, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - SZTE ÁOK Szent Györgyi Albert Klinikai Kozpont, Szeged
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Italy (8):
  - Casa di Cura Privata Malzoni - Villa dei Platani, Avellino, Campania
  - A.O.U. di Bologna Policlinico S.Orsola Malpighi, Bologna, Emilia-Romagna
  - A.S.U. Integrata di Udine, Udine, Friuli Venezia Giulia
  - Fondazione Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - IRCCS A.O.U. San Martino IST Ist. Nazionale Ricerca Cancro, Genoa, Liguria
  - A.O.U. Careggi, Florence, Tuscany
  - A.O.U. Senese, Siena, Tuscany
  - A.O.U. Integrata Verona, Verona, Veneto
- Netherlands (2):
  - Flevoziekenhuis, Almere Stad
  - Isala, Zwolle
- Poland (8):
  - CLINICAL MEDICAL RESEARCH Sp. z o. o., Katowice
  - Vita Longa Sp. z o.o., Katowice
  - Prywatny Gabinet Lekarski Ginekologia, Poloznictwo i Ultr., Lodz
  - Specjalistyczny Gabinet Ginekologiczno-Polozniczy, Lublin
  - NZOZ NOVITA, Specjalistyczne Gabinety Lekarskie, Lublin
  - VitroLive Sp. z o.o., Szczecin
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - NZOZ Zieniewicz Medical, Warsaw
- Spain (6):
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario "La Paz", Madrid
  - Hospital Regional de Málaga, Málaga
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital General Universitario de Valencia, Valencia
- United Kingdom (4):
  - York Teaching Hospital NHS Foundation Trust, York, North Yorkshire
  - Liverpool Womens Hospital, Liverpool
  - Norfolk and Norwich Hospital, Norwich
  - Whiston Hospital, Prescot

REFERENCES:
- [Derived] Hilpert J, Groettrup-Wolfers E, Kosturski H, Bennett L, Barnes CLK, Gude K, Gashaw I, Reif S, Steger-Hartmann T, Scheerans C, Solms A, Rottmann A, Mao G, Chapron C. Hepatotoxicity of AKR1C3 Inhibitor BAY1128688: Findings from an Early Terminated Phase IIa Trial for the Treatment of Endometriosis. Drugs R D. 2023 Sep;23(3):221-237. doi: 10.1007/s40268-023-00427-5. Epub 2023 Jul 9. PMID 37422772